CLINICAL TRIAL: NCT06327867
Title: Comparison of Video Laryngoscopy Versus Direct Laryngoscopy for Orotracheal Intubation Among Adults in Emergency Department
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Patan Academy of Health Sciences (Other)
Responsible Party: Principal Investigator, Rony Maharjan, Doctor, Lecturer, Department of General practice and Emergency medicine, Priniciple Investigator, Patan Academy of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: drs2402021836
Record Dates: First submitted 2024-03-18; First posted 2024-03-25 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: To Compare Success Rate of Video Laryngoscopy vs Direct Laryngoscopy
Keywords: Video Laryngoscope, Direct Laryngoscope

STUDY DESIGN:
Intervention Model Description: An open-label, single center, prospective, randomized, comparative, intervention study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Direct Laryngoscopy (Active Comparator): All participants who are intubated from Direct laryngoscopy is enrolled in this arm.
  Interventions: Device: Oro Tracheal Intubation by DL
- Video Laryngoscopy (Experimental): All participants who are intubated from Video laryngoscopy is enrolled in this arm.
  Interventions: Device: Oro Tracheal Intubation by VL

INTERVENTIONS:
Device: Oro Tracheal Intubation by DL — DL
  Arms: Direct Laryngoscopy
Device: Oro Tracheal Intubation by VL — VL
  Arms: Video Laryngoscopy

SUMMARY:
This is an open-label, single center, prospective, randomized, comparative, intervention study.

The goal of this study is to compare the success rate of video laryngoscopy vs direct laryngoscopy for first pass oro tracheal intubation. The other question it aims to answer are:

1. To assess the adverse events during video laryngoscopy
2. To assess the adverse events during direct Laryngoscopy
3. To compare the first pass success rate of DL vs VL according to demographic profile (age and sex)

DETAILED DESCRIPTION:
All consecutive patients presenting in Emergency medicine room requiring intubation, will be recruited in this study after taking informed written consent from the patients' family, excluding those falling in exclusion criteria. Direct laryngoscopy will be done by Mackintosh Laryngoscope with blade no 3 or 4. Video Laryngoscopy will be done by Mcgrath Mac Video Laryngoscope in respective groups. Intubations will be done by ER physicians and Emergency fellows of Emergency department. The total number of required sample size will be calculated and the obtained number will be divided in a group of 21 with block of 6 each. After randomizing the group and the block from a computerized software, a total of 21 envelope will be prepared in a consecutive manner and the patient will be intubated as per the pre decided blocks. All the patients in emergency who require intubation and falling into the inclusion criteria will be assessed. Informed written consent will be taken from the patient's family explaining that they will be a part of study and either of the laryngoscopy method will be used in them. Informed consent will be taken by one of the investigators, (ER physicians and emergency medicine fellow) who will be performing intubations in them.Inclusion criteria-

* Age 18 years
* Patient requiring orotracheal intubation
* Those who give written informed consent

Exclusion criteria-

* Pregnancy
* Intubations done by medical officers

Randomization-

* The consecutive patients will be assigned numbers serially from one.
* Block randomization of the patients in two arms will be done by using computerized software.

A total of 63 patients in each arm with total 126 patients will be included in the study. Blocks of 6 will be taken with total 21 groups. With using the software, random group will be selected and intubations will be done accordingly.

Demographic and clinical profile of patients in both arms will be recorded. Two treatment arms-

* Arm A- Orotracheal intubation done by Direct Laryngoscopy
* Arm B- Orotracheal intubation done by Video Laryngoscopy

Outcomes Primary- First pass success of direct laryngoscopy in oro tracheal intubation First pass success of video laryngoscopy in oro tracheal intubation

Secondary- Complications rates between two methods. Use of alternative methods for ventilation or oxygenation between two methods Better visualization of Cormack-Lehane grading between two methods

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years
2. Patient requiring orotracheal intubation
3. Those who give written informed consent

Exclusion Criteria:

1. Pregnancy
2. Intubations done by medical officers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
First pass success of direct laryngoscopy in oro tracheal intubation | 1 year
  success of oro tracheal intubation during DL
First pass success of video laryngoscopy in oro tracheal intubation | 1 year
  success of oro tracheal intubation during VL

SECONDARY OUTCOMES:
Complications rates between two methods. | 1 year
  rate of complication during intubation via DL or VL will be noted
Use of alternative methods for ventilation or oxygenation between two methods | 1 year
  use of alternative methods during intubation via DL or VL will be noted
Better visualization of Cormack-Lehane grading between two methods | 1 year
  better visualization of cormack lehane grading during intubation via DL or VL will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Rony Maharjan, MD, Principal Investigator — Patan Academy of Health Sciences

IPD SHARING:
Plan to Share IPD: No